CLINICAL TRIAL: NCT05902013
Title: Video Laryngoscopy Versus Direct Laryngoscopy for Nasotracheal Intubation in Neonates and Infants With Congenital Heart Disease Less Than 1-year of Age Prior Cardiac Surgery: a Pilot Study
Brief Title: Video Laryngoscopy Versus Direct Laryngoscopy for Nasotracheal Intubation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Eva M. Base, MD, PhD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11352022
Record Dates: First submitted 2023-05-21; First posted 2023-06-13 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Congenital Heart Disease; Airway Complication of Anesthesia
Keywords: Endotracheal intubation
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Laryngoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Video (Active Comparator): using video laryngoscopy for endotracheal intubation
  Interventions: Device: laryngoscopy
- Direct (Active Comparator): using direct laryngoscopy
  Interventions: Device: laryngoscopy

INTERVENTIONS:
Device: laryngoscopy — laryngoscopy for nasotracheal intubation

SUMMARY:
The aim of this study is to perform a pilot study investigating the first attempt intubation success rate differing between video laryngoscope nasotracheal intubation and direct laryngoscope nasotracheal intubation.

The study population will consist of 60 neonates and infants with congenital heart disease less than 1 year of age who need nasotracheal intubation during general anesthesia for cardiac procedures.

Standard nasotracheal intubation will be performed using either a video laryngoscope or direct laryngoscopy. Neonates and infants will be randomly assigned (1:1) to standard video laryngoscopy (with one of the following systems: Storz C-MAC Miller Video Laryngoscope, Karl Storz, Tuttlingen, Germany or Mc Grath Video Laryngoscope, Medtronic, Boulder,USA) or to direct laryngoscopy with one of the following blades: Miller or Macintosh (Heine, Hersching, Germany).

ELIGIBILITY:
Inclusion criteria.

* Age less than 1 year
* Congenital heart disease
* Scheduled for cardiac surgery
* Planned postoperative ICU stay

Exclusion criteria

* Nostrils not suitable for nasotracheal intubation
* Bleeding during dilation of nostrils

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
first attempt intubation success rate | study period, 30 minutes
  number

CONTACTS AND LOCATIONS:
Overall Officials: Eva M Base, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No